CLINICAL TRIAL: NCT03102359
Title: Cerebral Protection Effect of Selective Head Cooling and Dexmedetomidine in Patients Undergoing Liver Transplantation
Brief Title: Brain Protection Effect of Selective Head Cooling and Dexmedetomidine in Patients Undergoing Liver Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Huawei He, Postgraduate, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TJ-IRB20170201
Record Dates: First submitted 2017-03-24; First posted 2017-04-05 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Liver Transplant; Complications
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Selective Head Cooling (Experimental): Participants received a cooling helmet filled with ice water mixture after an-esthesia induction until the end of the surgery.
  Interventions: Device: Cooling Helmet
- Dexmedetomidine (Experimental): Giving dexmedetomidine1μg/kg i.v for 10 minutes, then use computerized infusion pump at 0.5μg/kg.h until the end of the surgery.
  Interventions: Drug: Dexmedetomidine
- Selective Head Cooling and Dexmedetomidine (Experimental): Using selective head cooling combined with dexmedetomidine as described before
  Interventions: Drug: Dexmedetomidine; Device: Cooling Helmet
- Control (No Intervention): No intervention in this group

INTERVENTIONS:
Drug: Dexmedetomidine — Using dexmedetomidine at anesthesia induction and maintain until the end of the surgery
  Arms: Dexmedetomidine; Selective Head Cooling and Dexmedetomidine
Device: Cooling Helmet — Using cooling helmet for selective head cooling group and Selective Head Cooling and Dexmedetomidine group
  Arms: Selective Head Cooling; Selective Head Cooling and Dexmedetomidine

SUMMARY:
The investigators investigated in the present study whether selective head cooling and dexmedetomidine has an effect on cerebral oxygenation during liver transplantation and has cerebral protective effect in patients undergoing liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for OLT, selected from the Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, China.
* Sign the informed consent

Exclusion Criteria:

* The patients with a history of neurological or psychiatric disorders which impair cognitive processes, including previously established de-mentia, stroke, schizophrenia and depression were excluded from the study.
* Patients diagnosed with hepatic encephalopathy or had a low Mini-Mental State Examination (MMSE) score (below 24) preoperatively.
* With concurrent diseases such as renal insufficiency, diabetes mellitus were also excluded.
* Patients were excluded if severe reperfusion syn-drome (mean arterial pressure below 60mmHg sustained over 15minutes) occurred perioperatively.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative minimal hepatic encephalopathy (MHE) | 14 days after surgery
  Using PSE-Syndrom-Test

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital,Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No